CLINICAL TRIAL: NCT00207025
Title: A Phase I Study of BMS-275183 Given on a Daily Schedule in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA165-012
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-07

CONDITIONS: Tumors
Keywords: Patients with advanced solid tumors
MeSH Terms: conditions — Neoplasms | interventions — BMS-275183

INTERVENTIONS:
Drug: BMS-275183

SUMMARY:
The purpose of this clinical research study is to learn about the safety and tolerability of daily BMS-275183 in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Non-hematologic malignancy that has progressed or no standard therapy is known
* Four weeks from last chemotherapy or two weeks from last non-cytotoxic therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* No more than 3 prior chemotherapy regimens in advanced/metastatic setting
* Absolute neutrophil count >=1,500/mm3 and platelets >=100,000/mm3
* Bilirubin <=1.5 x Upper Limit of Normal (ULN), Aspartate aminotransferase <=2.5 x ULN
* Serum creatinine <=1.5 x ULN
* Men and women >=18 years
* Women of Child Bearing Potential (WOCBP) must use adequate method of contraception throughout and up to 4 weeks after the study

Exclusion Criteria:

* WOCBP and men not using adequate method of birth control
* WOCBP who are pregnant or breastfeeding
* Prior radiation >=25% of bone marrow containing skeleton
* Uncontrolled, significant, or active cardiovascular or pulmonary disease or infection or psychiatric disorder
* Neuropathy
* Active brain metastases
* Inability to swallow capsules
* History of gastrointestinal disease, surgery or malabsorption, or requiring use of a feeding tube
* Concurrent chemotherapy, hormonal therapy, immunotherapy, or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability

SECONDARY OUTCOMES:
PK, preliminary evidence of antitumor activity

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Local Institution, Detroit, Michigan
  - Local Institution, Pittsburgh, Pennsylvania
- Local Institution, Brussels, Belgium